CLINICAL TRIAL: NCT07253467
Title: Load Dependent Modulation of Spinal Excitability: Linking H-Reflex Supression and Whole Body Vibration Induced Reflex Latency
Acronym: SRML
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, İsmet Alkım Özkan, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IstPRMTRH2A
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Vibration; H-reflex
Keywords: H-Reflex; Whole Body Vibration; Bone Myoregulation Reflex; Reflex Latency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy participants (Experimental): Participants will complete a series of experimental tasks involving postural mechanical and vibrational loading. The protocol consists of quiet standing on both feet, single-leg standing on the left side, standing during whole-body vibration (WBV), and single-leg standing on the left side during WBV. Vibration amplitudes of 2.2 mm and 1.2 mm will be applied in each condition. H-reflex measurements will be recorded from the soleus muscle throughout all tasks to evaluate alterations in spinal reflex excitability. Vibration induced reflex latency will be also measured with different vibration frequencies (30-32-34-36) also measured in the same protocol.
  Interventions: Other: Whole Body Vibration

INTERVENTIONS:
Other: Whole Body Vibration — Whole Body Vibration (WBV) is a neuromuscular training modality in which patients stand, sit, or exercise on a platform that delivers mechanical oscillations (30-36 Hz, 1-2 mm amplitude). While WBV is applied H-Reflex tests are done.

SUMMARY:
This study examines how different standing postures and whole-body vibration conditions affect spinal reflex activity. Participants will stand in various positions-with and without vibration of two amplitudes-and H-reflex responses from the soleus muscle will be recorded. Additionally, vibration-induced reflex latency will be assessed across multiple vibration frequencies.

DETAILED DESCRIPTION:
Participants will engage in a structured set of experimental tasks designed to evaluate the effects of postural mechanical loading, and whole-body vibration.

The protocol includes four primary standing conditions:

Quiet bipedal stance,

Single-leg stance on the left side,

Bipedal stance during whole-body vibration (WBV), and

Single-leg stance on the left side during WBV.

During all WBV conditions, two vibration amplitudes-2.2 mm and 1.2 mm-will be applied sequentially to assess amplitude-dependent modulation of reflex responses.

Throughout each condition, H-reflex recordings from the soleus muscle will be collected to quantify changes in spinal reflex excitability under varying postural and vibratory loads. In addition to these measurements, vibration-induced reflex latency will be evaluated by delivering vibratory stimuli at multiple frequencies (30, 32, 34, and 36 Hz) within the same experimental protocol. This approach allows for a comprehensive analysis of how both posture and vibratory parameters influence neuromuscular reflex pathways.

The investigators conducted an a priori power analysis for a repeated-measures ANOVA (within-subjects design) to determine the required sample size. The analysis was based on a medium expected effect size, specified as partial eta squared (ηₚ²) = 0.06, which corresponds to an effect size of f = 0.25. The investigators set the alpha error probability at 0.05 and the desired statistical power (1-β) at 0.80. The design included one group with five repeated measurements, assuming a correlation of 0.70 among repeated measures. Under these conditions, the critical F value was 2.5652405, with 4 numerator degrees of freedom and 48 denominator degrees of freedom. The power analysis indicated that a total sample size of 13 participants is required. The required sample size was calculated using G*Power version 3.1.9.4 (Franz Faul, University of Kiel, Germany).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between 25 and 50 years of age
* Individuals willing to participate and able to provide informed consent
* Individuals who can stand independently for at least 10 minutes
* Participants with no known neurological, orthopedic, or balance impairments

Exclusion Criteria:

* Individuals who can not tolerate WBV
* Individuals who can not tolerate electrical stimulation
* Pregnancy

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2025-12-08 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Whole Body Vibration induced reflex latency | Day 1 (single-session, during each experimental condition)
  WBV induced reflex latency will be measured
H-Reflex Size | Day 1 (single-session, during each experimental condition)
  Peak to peak amplitude of the H-Reflex will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Bahçelievler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes